CLINICAL TRIAL: NCT06033430
Title: The Effectiveness of Dry Needling in Treating Linear Hypertrophic Scar Tissue: a Randomized Sham-controlled Trial
Brief Title: Effectiveness of Dry Needling in Linear Scar Tissue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.IUMS.REC.1401.540
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-11

CONDITIONS: Scar Tissue; Hypertrophic Scar; Hypertrophic Scar of Upper Arm (Disorder); Hypertrophic Surgical Scar; Dry Needling
Keywords: Hypertrophic scar; Dry needling; Randomized sham-controlled trial
MeSH Terms: conditions — Cicatrix; Cicatrix, Hypertrophic

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the control group will undergo the same procedure as those in the intervention group, with needles placed superficially in an area slightly further away from the scar tissue. Furthermore, to minimize bias, the data analyst will be blinded to the grouping of the participants, and each participant will be identified by a unique numerical code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True dry needling of the hypertrophic scar tissue (Experimental): Participants with hypertrophic linear scar tissue in the true dry needling group will undergo authentic dry needling interventions targeted at the scar tissue, in conjunction with routine physiotherapy.
  Interventions: Other: True dry needling
- Sham dry needling of the hypertrophic scar tissue (Sham Comparator): In the sham dry needling group, participants presenting with hypertrophic linear scar tissue will receive superficial dry needling of the skin, performed at a location distinct from the scar tissue. This will be administered alongside routine physiotherapy.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Other: True dry needling — Prior to the procedure, participants will be given a detailed explanation of the dry needling technique. Afterward, the specific area will be thoroughly cleaned using an alcohol pad. In the true dry needling group, along with routine physiotherapy, a sterile filiform acupuncture needle, measuring 2 cm in length and designed for single-use, will be inserted at a 15-degree angle relative to the skin's surface, directly into the scar tissue. Once inserted, the needle will be gently rotated to aid in separating tissue adhesions along the path of the scar. Routine physiotherapy includes the application of kinesiology taping, in addition to a 20-minute session of infrared therapy positioned 30 cm away from the scar tissue. A total of six treatment sessions will be administered to the patients, with three sessions per week scheduled over a two-week period.
  Arms: True dry needling of the hypertrophic scar tissue
Other: Sham dry needling — The sham group participants will be positioned in a similar manner to those in the experimental group, with a minor exception. Instead of inserting the 2-cm single-use sterile filiform acupuncture needle into the scar tissue, it will be superficially inserted at a point further away from the scar tissue and removed after 20 minutes. Moreover, routine physiotherapy administered to the participants in the sham group will be identical to that of the experimental group, ensuring consistency between the two groups.
  Arms: Sham dry needling of the hypertrophic scar tissue

SUMMARY:
Scar tissue can cause serious complications that significantly impact a patient's quality of life. Common complications include stiffness and contractions, which can restrict joint mobility and make daily activities challenging. In severe cases, these limitations can even prevent patients from fulfilling their work responsibilities or engaging in activities they enjoy. The deleterious effect of scar tissue on a patient's well-being is of utmost significance. However, several therapeutic approaches have been proposed to manage scar tissue complications. Enhancing scar tissue compliance can help patients regain their functional abilities and reduce limitations. One such approach is dry needling, a technique used to improve the flexibility of myofascial tightness. Nevertheless, the effectiveness of dry needling in improving scar tissue compliance remains debatable. Therefore, this study aims to investigate the therapeutic effects of dry needling on complications resulting from linear hypertrophic scars caused by surgery or trauma.

DETAILED DESCRIPTION:
RESEARCH OBJECTIVE:

The primary objective of this study is to investigate the effectiveness of dry needling on hypertrophic scar tissue compliance using a compliance meter. The secondary objectives of the study are to evaluate active and passive range of motion, pain, and functional disability.

RESEARCH DESIGN:

This study is a two-centered, randomized, single-blind, sham-controlled trial with an allocation ratio of 1:1. Eighty participants with hypertrophic scar tissue will be randomly assigned into two groups with equal sample size. Random allocation will be performed using the permuted block randomization method, consisting of four-letter blocks made of letters A and B. The random treatment list obtained at the end of the random allocation task will be placed in letters A and B inside sealed and numbered envelopes. The random assignment process will be performed by someone outside the research team before the study begins.

PROCEDURE:

Eligible participants will be asked to complete an intake form providing demographic data such as age, gender, height, weight, occupation, and questions related to their scar tissue (onset, injury mechanism, location, duration, and whether it causes pain). The principal investigator will confirm each participant's eligibility. Next, each participant will complete a pain and functional disability questionnaire. After gathering subjective information, tissue compliance data and active and passive range of motion near the nearest joint next to the scar tissue will be collected. The outcome measurements will be administered in an order of tissue compliance, followed by joint active and passive range of motion.

INTERVENTION:

After the baseline assessment, the principal investigator will administer the dry needling intervention. For the intervention group, a 2-cm sterile, disposable, solid filament needle (Dongbang Acupuncture Needle, Korea) will be manually inserted at an angle of approximately 15 degrees to the skin surface into the scar tissue. The needle will then be rotated to separate the tissue adhesions along the path of the scar tissue. In the sham dry needling treatment group, the patient's condition will be identical to that of the real dry needling treatment group, with a minor exception. Instead of inserting the 2-cm single-use sterile filiform acupuncture needle into the scar tissue, it will be superficially inserted at a point further away from the scar tissue and removed after 20 minutes. Both groups will receive basic routine treatment, including kinesiology taping, along with infrared therapy (for 20 minutes) at a distance of 30 cm from the scar tissue. The patients will undergo six treatment sessions, with three sessions per week for two weeks.

REASSESSMENT:

After the interventions, measures of the primary and secondary outcomes will be collected immediately and two weeks after the final treatment session to evaluate the effectiveness of the dry needling intervention. Additionally, any adverse events following the dry needling procedures will be assessed immediately, such as bruising, nausea, dizziness, or post-needling soreness. If bleeding occurs, the participant will be informed.

ELIGIBILITY:
Inclusion Criteria:

* Linear hypertrophic scar tissue with an age of more than six weeks
* No restrictions on active and passive joint range of motion near the scar tissue
* Age between 20 and 60 years

Exclusion Criteria:

* Needle phobia
* Immature scar or keloid scar
* Skin diseases or infections near the scar tissue
* Diabetes
* Fractures that have altered joint mobility
* Anticoagulant medication use

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Flexibility of the scar tissue (tissue compliance) | Change in flexibility of the scar tissue after the end of 6 treatment sessions compared to baseline and change from baseline at 2-week follow up
  The Tissue Compliance Meter (STCM), created by the Technical University of Chemnitz in Germany, is a straightforward tool for measuring tissue compliance. It consists of a ruler with millimeter markings, attached to a standard algometer from Greenwich, CT, USA. It also includes two additional components: a round plastic disk with a metal cylinder and a ring with a screw for securing them in place. These disk and ring components can be adjusted along the ruler. A button cell battery is used to generate a beep when the ring and disk touch each other. To take a measurement, the investigator pushes the top of the algometer into the tissue until it reaches displacements of 0.5, 1, and 1.5 centimeters on the scar tissue. The investigator then records the applied force in either kilograms or Newtons, depending on the pre-set displacement. Each measurement is repeated three times, and the average of these three repetitions is used for statistical analysis.

SECONDARY OUTCOMES:
Active and passive joint range of motion | Change in joint range of motion after the end of 6 treatment sessions compared to baseline and change from baseline at 2-week follow up
  To assess joint active and passive range of motion, a 360-degree universal goniometer will be used. This involves correctly positioning and stabilizing the joint, moving the body part through its appropriate range of motion, determining the joint's end of the range and its end-feel, palpating the relevant bony landmarks, aligning the goniometer with these landmarks, and accurately reading the measuring instrument. Each measurement will be repeated three times, and the average of these repetitions will be used for statistical analysis.
Pain intensity | Change in pain after the end of 6 treatment sessions compared to baseline and change from baseline at 2-week follow up
  If pain is present in the scar region, the Numeric Pain Rating Scale (NPRS) will be employed to assess pain intensity. This scale, ranging from 0 (indicating no pain) to 10 (representing the most severe pain imaginable), will be used for rating by participants during the evaluation. The NPRS is a pain assessment tool commonly utilized in research. In this study, a minimum clinically significant difference of 0.2 will be considered.
Health-related quality of life | Change in health status after the end of 6 treatment sessions compared to baseline and change from baseline at 2-week follow up
  Following dry needling, the assessment of health status will be conducted using the SF-36 questionnaire, which includes 36 questions related to an individual's quality of life. This evaluation produces two summary scores: one for physical health and another for mental health.

CONTACTS AND LOCATIONS:
Locations (2):
- Myopain Seminars, Bethesda, Maryland, United States
- School of Rehabilitation Sciences, Iran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
The data sets of this study will be available on a reasonable request to the corresponding author.
Time Frame: Starting 6 months after the publication.

REFERENCES:
- [Background] Alaei P, Nakhostin Ansari N, Naghdi S, Fakhari Z, Komesh S, Dommerholt J. Dry Needling for Hamstring Flexibility: A Single-Blind Randomized Controlled Trial. J Sport Rehabil. 2020 Oct 7;30(3):452-457. doi: 10.1123/jsr.2020-0111. PMID 33027765
- [Background] Bartsch K, Brandl A, Weber P, Wilke J, Bensamoun SF, Bauermeister W, Klingler W, Schleip R. Assessing reliability and validity of different stiffness measurement tools on a multi-layered phantom tissue model. Sci Rep. 2023 Jan 16;13(1):815. doi: 10.1038/s41598-023-27742-w. PMID 36646734
- [Background] Gandbhir VN, Cunha B. Goniometer. 2020 Jun 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK558985/ PMID 32644411
- [Background] Lubczynska A, Garncarczyk A, Wcislo-Dziadecka D. Effectiveness of various methods of manual scar therapy. Skin Res Technol. 2023 Mar;29(3):e13272. doi: 10.1111/srt.13272. PMID 36973982
- [Background] Bahramian M, Dabbaghipour N, Aria A, Sajadi Moghadam Fard Tehrani B, Dommerholt J. Efficacy of Dry Needling in Treating Scars following Total Hip Arthroplasty: A Case Report. Med J Islam Repub Iran. 2022 Dec 20;36:156. doi: 10.47176/mjiri.36.156. eCollection 2022. PMID 36660004
- [Background] Rozenfeld E, Sapoznikov Sebakhutu E, Krieger Y, Kalichman L. Dry needling for scar treatment. Acupunct Med. 2020 Dec;38(6):435-439. doi: 10.1177/0964528420912255. Epub 2020 Mar 30. PMID 32228036
- [Background] Deflorin C, Hohenauer E, Stoop R, van Daele U, Clijsen R, Taeymans J. Physical Management of Scar Tissue: A Systematic Review and Meta-Analysis. J Altern Complement Med. 2020 Oct;26(10):854-865. doi: 10.1089/acm.2020.0109. Epub 2020 Jun 24. PMID 32589450
- [Background] Tanaka Y, Matsuo K, Yuzuriha S. Long-term histological comparison between near-infrared irradiated skin and scar tissues. Clin Cosmet Investig Dermatol. 2010 Nov 25;3:143-9. doi: 10.2147/CCID.S15729. PMID 21437069
- [Background] Kurtti A, Nguyen JK, Weedon J, Mamalis A, Lai Y, Masub N, Geisler A, Siegel DM, Jagdeo JR. Light emitting diode-red light for reduction of post-surgical scarring: Results from a dose-ranging, split-face, randomized controlled trial. J Biophotonics. 2021 Jul;14(7):e202100073. doi: 10.1002/jbio.202100073. Epub 2021 May 4. PMID 33788987
- [Background] Klingenstein A, Garip-Kuebler A, Muth DR, Hintschich C. A prospective randomized pilot study evaluating the scar outcome after gluteal dermis fat graft with and without kinesiotaping. Int Ophthalmol. 2022 Aug;42(8):2563-2571. doi: 10.1007/s10792-022-02304-7. Epub 2022 Apr 2. PMID 35366138
- [Background] O'Reilly S, Crofton E, Brown J, Strong J, Ziviani J. Use of tape for the management of hypertrophic scar development: A comprehensive review. Scars Burn Heal. 2021 Jul 12;7:20595131211029206. doi: 10.1177/20595131211029206. eCollection 2021 Jan-Dec. PMID 34290886
- See also: Related Info — https://www.thysol.us/kinesiology-tape-instructions/scars/
- See also: Related Info — https://apta.confex.com/apta/csm2020/meetingapp.cgi/Paper/21253